CLINICAL TRIAL: NCT00134017
Title: HLA Matched Related and Unrelated Bone Marrow Transplantation With Busulfan/Cyclophosphamide and Post Transplantation Cyclophosphamide for Hematological Malignancies
Brief Title: Combination Chemotherapy, Bone Marrow Transplant, and Post Transplant Cyclophosphamide for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0373; P01CA015396 (NIH); P30CA006973 (NIH); NA_00034100 (Other: JHMIRB)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia in remission; refractory anemia with excess blasts; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage II multiple myeloma; stage III multiple myeloma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; chronic myelomonocytic leukemia; refractory chronic lymphocytic leukemia; refractory multiple myeloma; secondary myelodysplastic syndromes; stage IV adult lymphoblastic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Hodgkin Disease; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Recurrence; Leukemia, Myelomonocytic, Chronic | interventions — Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: US Export: No

ARMS (1):
- Bone marrow transplant (Experimental): Myeloablative bone marrow transplant with a busulfan (Bu), cyclophosphamide (Cy), preparative regimen and post-transplant cyclophosphamide (PTCy) as GVHD prophylaxis
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Busulfan — Days -7 to -4: 4 mg/kg PO daily OR 3.2 mg/kg IV daily OR 160 mg/m^2 daily (for pediatric recipients)
  Other Names: Myleran; Busulfex
Drug: Cyclophosphamide — Days -3, -2, +3, +4: 50 mg/kg IV daily
  Other Names: Cytoxan; CTX

SUMMARY:
RATIONALE: Giving chemotherapy before a donor bone marrow transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclophosphamide, mycophenolate mofetil, or tacrolimus after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with tacrolimus and mycophenolate mofetil works in treating patients who are undergoing a donor bone marrow transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the optimal dose of post-transplant immunosuppression comprising high-dose cyclophosphamide, tacrolimus, and mycophenolate mofetil administered after myeloablative conditioning chemotherapy comprising busulfan and cyclophosphamide followed by allogeneic bone marrow transplantation in patients with high-risk hematologic malignancies.
* Determine the incidence and severity of acute graft-versus-host disease in patients treated with this regimen.
* Determine other toxic effects of this regimen in these patients.

Secondary

* Determine immune reconstitution in patients treated with this regimen.
* Determine disease control in patients treated with this regimen.

OUTLINE: This is a pilot study. Patients are stratified according to age (≤ 19 years old vs > 19 years old).

* Myeloablative conditioning chemotherapy: Patients receive busulfan IV or orally 4 times daily on days -7 to -4 OR days -6 to -3 and cyclophosphamide IV over 1 hour once daily on days -3 to -1 OR days -2 and -1.
* Allogeneic bone marrow transplantation: Patients undergo allogeneic bone marrow transplantation on day 0.
* Immunosuppression therapy: Patients receive high-dose cyclophosphamide IV over 1 hour on days 3 and 4.

After completion of study transplantation, patients are followed at 30 and 60 days, 6 months, 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * AML beyond first complete remission (CR1)
    * Refractory AML
    * AML arising from myelodysplastic syndromes (MDS)
    * Secondary AML
  * MDS

    * Refractory anemia with excess blasts with > 10% blasts in bone marrow
  * Acute lymphoblastic leukemia (ALL), meeting 1 of the following criteria:

    * ALL in CR1 with 1 of the following high-risk features:

      * Philadelphia chromosome (Ph)-positive disease
      * Less than 1 year of age at diagnosis
      * Cytogenetic abnormalities involving chromosome 11q23
    * ALL beyond CR1
    * Refractory ALL
  * Chronic myeloid leukemia beyond first chronic phase
  * Chronic myelomonocytic leukemia
  * Chronic lymphocytic leukemia

    * Stage III-IV disease
    * Does not meet criteria for other bone marrow transplantation (BMT) studies
  * Myeloproliferative disorders

    * Ph-negative disease
  * Hodgkin's or non-Hodgkin's lymphoma

    * Chemotherapy-resistant disease
  * Paroxysmal nocturnal hemoglobinuria with life-threatening thrombosis
  * Multiple myeloma

    * Stage II or III disease
* Very high-risk disease

  * Having an unrelated donor is considered a high-risk condition
* Meets medical criteria for myeloablative BMT for the Sidney Kimmel Comprehensive Cancer Center
* Bone marrow donor available, meeting 1 of the following criteria:

  * Genotypically HLA-identical sibling
  * Phenotypically matched first-degree relative
  * Unrelated donor molecularly matched at HLA-A, -B, -C, -DRB1, and -DQB1

PATIENT CHARACTERISTICS:

Age

* 6 months to 65 years

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* No concurrent dexamethasone as an antiemetic during immunosuppression therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent immunosuppressants until ≥ 24 hours after the completion of cyclophosphamide (post-transplantation)

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Luznik, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luznik L, Bolanos-Meade J, Zahurak M, Chen AR, Smith BD, Brodsky R, Huff CA, Borrello I, Matsui W, Powell JD, Kasamon Y, Goodman SN, Hess A, Levitsky HI, Ambinder RF, Jones RJ, Fuchs EJ. High-dose cyclophosphamide as single-agent, short-course prophylaxis of graft-versus-host disease. Blood. 2010 Apr 22;115(16):3224-30. doi: 10.1182/blood-2009-11-251595. Epub 2010 Feb 2. PMID 20124511

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Marrow Transplant
Started | 142
Completed | 142
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 123
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 47 [21 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Develop Acute Graft-versus-host Disease (GVHD)
Description: Percentage of participants who developed grades II-IV and grades III-IV acute GVHD. Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade I (skin involvement stages 1+ to 2+, with no liver or GI involvement), Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+).
Time Frame: Day 100
Population: The study data was analyzed early after 117 participants had been treated. This was done in order to publish the data and establish a new local standard of care at our institution. GVHD data was collected on 15 additional participants for a total of 132. GVHD data was not collected on the remaining 10 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 132
Participants
  Grades II-IV acute GVHD | 49
  Grades III-IV acute GVHD | 10

2. Secondary Outcome: Days to Engraftment
Description: Median number of days to neutrophil and platelet engraftment.
Time Frame: Up to one year
Population: The study data was analyzed early after 117 participants had been treated. This was done in order to publish the data and establish a new local standard of care at our institution. Engraftment data was not collected on the remaining 25 participants. Recipients of related-donor (n=78) and unrelated-donor (n=39) transplants were reported separately.
Measure: Median (Full Range); unit: days
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 117
days
  Neutrophil engraftment, related donors: number analyzed (Participants) | 78
  Neutrophil engraftment, related donors | 23 [2 to 100]
  Neutrophil engraftment, unrelated donors: number analyzed (Participants) | 39
  Neutrophil engraftment, unrelated donors | 25 [2 to 100]
  Platelet engraftment, related donors: number analyzed (Participants) | 78
  Platelet engraftment, related donors | 31 [5 to 354]
  Platelet engraftment, unrelated donors: number analyzed (Participants) | 39
  Platelet engraftment, unrelated donors | 35 [5 to 354]

3. Secondary Outcome: Chimerism
Description: Number of patients who achieved 100% donor chimerism.
Time Frame: Day 30, Day 60
Population: The study data was analyzed early after 117 participants had been treated. This was done in order to publish the data and establish a new local standard of care at our institution. Chimerism data was not collected on the remaining 25 participants. One participant died prior to Day 30 and was not analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 116
Participants
  Day 30 | 99
  Day 60 | 101

4. Secondary Outcome: Non-relapse Mortality
Description: Percentage of participants who died for BMT-related reasons.
Time Frame: Day 100, 2 years
Population: The study data was analyzed early after 117 participants had been treated. This was done in order to publish the data and establish a new local standard of care at our institution. NRM data was not collected on the remaining 25 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 117
percentage of participants
  Day 100 | 6 [2 to 13]
  2 years | 15 [8 to 24]

5. Secondary Outcome: Relapse
Description: Percentage of participants who developed relapse or progressive disease.
Time Frame: 2 years
Population: The study data was analyzed early after 117 participants had been treated. This was done in order to publish the data and establish a new local standard of care at our institution. Relapse data was not collected on the remaining 25 participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bone Marrow Transplant
Number analyzed (Participants) | 117
percentage of participants | 44 [34 to 53]

ADVERSE EVENTS:
Time Frame: Up to one year
Description: Adverse events were tracked systematically for 30-60 days depending on exact discharge date from the initial hospitalization.
  Only the following adverse events were collected: all graft failures; deaths in the first sixty days; unexpected grade 4-5 events.
Arm/Group | Bone Marrow Transplant
All-Cause Mortality (participants affected / at risk) | 66/142
Serious Adverse Events (participants affected / at risk) | 20/142
Other Adverse Events (participants affected / at risk) | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplant (N=142)
Aspergillus pneumonia (Infections and infestations) | 1 (1)
Graft failure (Immune system disorders) | 6 (6)
Graft versus host disease (Immune system disorders) | 1 (1)
Multiorgan failure (Immune system disorders) | 1 (1)
Pulmonary failure (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Veno-occlusive disease (Hepatobiliary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes